CLINICAL TRIAL: NCT04419584
Title: A Randomized Placebo-Controlled Clinical Trial of an Innovative Herbal Formula for Atopic Dermatitis in Children: Evaluations of Modified Qing-Ying Decoction on Efficacy and Gut Microbiome
Brief Title: Evaluate the Efficacy of Using Modified Qing-Ying Decoction in Atopic Dermatitis Children
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Associate professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD study
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Qing-Ying Decoction (Experimental): Herbal granules, twice per day for 12 weeks
  Interventions: Drug: Modified Qing-Ying Decoction
- Identical looking placebo (Placebo Comparator): Placebo granules, twice per day for 12 weeks
  Interventions: Drug: Identical looking placebo

INTERVENTIONS:
Drug: Modified Qing-Ying Decoction — Herbal granules
  Arms: Modified Qing-Ying Decoction
Drug: Identical looking placebo — Placebo granules
  Arms: Identical looking placebo

SUMMARY:
The study aims to evaluate the clinical efficacy and safety of the modified Qing-Ying Decoction (mQYD) for the treatment of subacute and chronic atopic dermatitis (AD) in children when compared to the placebo control through examining the clinical symptoms, quality of life, gut microbiome, and Chinese medicine body constitution.

This is a parallel, randomized, placebo-controlled, double-blind clinical trial. Eligible subjects will be randomly allocated to receive oral mQYD granules or it's placebo granules. Subjects will have 12-week of treatment, and then a 4-week follow-up.

DETAILED DESCRIPTION:
The subjects will come for a screening visit at week 0 (baseline), then at week 6, week 12, and week 16 for Chinese medicine practitioner (CMP) investigators assessments. Eczema Area and Severity Index (EASI), Children's Dermatology Life Quality Index (CDLQI), Patient-Oriented Eczema Measure (POEM), and Chinese Medicine body constitution types will be assessed and filled up at different timepoints. They will receive oral herbal mQYD or placebo granules for 12 weeks and then be followed up 4 weeks after the treatment. Registered CMPs will provide consultation under Chinese medicine theory. Study medication compliance and adverse events will also be assessed at each visit. Besides, they need to record the food taken in a diary before the day for taking faecal specimen for gut microbiome analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 4 to 17 (Chinese only);
2. With EASI ≥ 10;
3. Subacute and chronic atopic dermatitis presenting with dry, scaly, erythematous papules and plaques; and
4. Provide written informed consent form (signed by one of their parents)

Exclusion Criteria:

1. History of allergy to Chinese medicines;
2. AD with Yang deficiency in syndrome differentiation, such as pale looking, always feeling cold, fatigue, chronic diarrhea with loose stool, urinary disorders such as urinary difficulty, excessive urination or incontinence
3. Known overt bacterial infections in the skin;
4. Known pregnancy;
5. Known severe medical conditions, such as cardiovascular, liver or renal dysfunction or Diabetes Mellitus;
6. Having used oral corticosteroids, oral antibiotics, other immunosuppressive or any preparation of oral herbal medicines for the treatment of AD in the past month;
7. Having been diagnosed with scabies, allergic contact dermatitis, seborrheic dermatitis or psoriasis; and
8. Has taken anti-coagulant or anti-platelet drugs in the past month.
9. Has taken any probiotics, prebiotics in the last month
10. Known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | 16 weeks
  Min value: 0, max value: 72, higher scores mean worse outcome. To assess the severity of atopic dermatitis

SECONDARY OUTCOMES:
Patient Oriented Eczema Measure (POEM) | 16 weeks
  Min value: 0, max value: 28, higher scores mean worse outcome. To assess the subjective symptoms of subjects.
Children's Dermatology Life Quality Index (CDLQI) | 16 weeks
  Min value: 0, max value: 30, higher scores mean worse outcome. To assess the quality of life of subjects.
Constitution of Chinese Medicine Questionnaire (CCMQ) | 16 weeks
  Not a scale. Based on the answers, a logarithm will be used to determine the type of Chinese Medicine Constitution of the subjects. To assess the Chinese medicine body constitution of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-xiu Lin, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No